CLINICAL TRIAL: NCT03304236
Title: Motion Analysis of the Myelopathy Hand: New Insight Into the Classical Sign
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 17-174
Record Dates: First submitted 2017-09-27; First posted 2017-10-06 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Cervical Myelopathy
Keywords: Cervical Myelopathy; sEMG; Motion capture analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myelopathy hand: Patients will undergo radiological and clinical examination at the Duchess of Kent Children Hospital. Patients will be required to put on a pair of hand gloves with 18 IMUs located on specific bony landmarks (distal phalanges of fingers, proximal phalanges of index fingers and thumbs, dorsum of the hands and bilateral wrists).
  Interventions: Device: Myelopathy Hand

INTERVENTIONS:
Device: Myelopathy Hand — Patients will undergo radiological and clinical examination at the Duchess of Kent Children Hospital. Patients will be required to put on a pair of hand gloves with 18 IMUs located on specific bony landmarks (distal phalanges of fingers, proximal phalanges of index fingers and thumbs, dorsum of the hands and bilateral wrists)

SUMMARY:
This study aims to quantify the clumsiness and decreased dexterity seen in the grip and release test using a simple glove with sensors that can quantify the abnormal motion of this classical sign. This new tool will give a mechanistic insight into the myelopathy. The findings of this study will also form the basis of a prospective longitudinal study with clinical and radiological evaluation to compare the prognosticating value of this new information in clinical practice.

DETAILED DESCRIPTION:
Cervical myelopathy is a common condition due to degeneration of the cervical spine causing stenosis and cord compression, with a higher prevalence in Asian population. It leads to decreased hand dexterity and function, sensory loss, gait and sphincter disturbance. Natural history shows a stepwise deterioration in most cases, whilst a slow progressive deterioration or sudden deterioration is observed in small number of subjects.

The myelopathy hand was first described by Ono et al. on the analysis of finger motion impairment caused by cervical myelopathy. They described a 10 second grip and release test, which documents the number of times a subject can make a fist and release it as rapidly as possible within 10 seconds. The clumsiness associated with intrinsic finger weakness decreases the number of cycles a patient can perform during the test. They quantified patients' neurologic deficit and found that <20 grip -release cycles in 10 seconds represented symptomatic myelopathy. The presence of this sign is not only pathognomonic of cervical myelopathy but also correlates with disease severity. This is a sensitive and specific sign of pyramidal tract involvement and has since become a classical sign and objective test of the condition. The presence of myelopathic hand signs aids the diagnosis of symptomatic cervical myelopathy and its grading acts a guide to the severity of the condition to the treating surgeon.

However, this quantitative analysis only provides a crude representation of the clumsiness that patients experience from their deterioration of hand function. In the original description, Ono et al. noted the quality of this movement was affected particularly in advanced cases, where there was difficult, slow and incomplete finger extension, exaggerated wrist flexion with attempted finger extension and exaggerated wrist extension with finger flexion. This was considered to be caused by a failure of synergy between the wrist and the fingers. Finger motion is complex, varies greatly and clinical evaluation is often difficult. Apart from the counting the number of cycles a patient can perform, the classical grip and release test contains other critical clinical information that has been widely described by surgeons but in very vague terms that are neither reproducible nor meaningful in clinical practice. Although this uncoordinated finger motion and inability to move their fingers smoothly in grip and release cycles are well-known phenomena in myelopathy patients, they have been only vaguely recognized. Presently these kinematic characteristics have not been quantified or studied, and it is not known which types of myelopathy present with them, how it correlates with disease severity and its prognosticating value.

ELIGIBILITY:
Inclusion Criteria:

* All degenerative causes of documented cervical myelopathy planned for operation will be recruited into the study.

Exclusion Criteria:

* Patients found to have spinal tumour, infection, or other non-degenerative causes as well as patient who are unable to follow command and/or unwilling to attend follow up will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at the Duchess of Kent Children's Hospital will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Objective quantification of the hand movement during grip and release test using sEMG and motion capture analysis | 1 year
  Objective quantification of the hand movement during grip and release test using sEMG and motion capture analysis

SECONDARY OUTCOMES:
Correlate the clinical severity of myelopathy with different patterns of hand movement using sEMG and motion capture analysis | 1 year
  To correlate the clinical severity of myelopathy with different patterns of hand movement using sEMG and motion capture analysis
Correlate the radiological level of myelopathy involvement with different patterns of hand movement using sEMG and motion capture analysis | 1 year
  To correlate the radiological level of myelopathy involvement with different patterns of hand movement using sEMG and motion capture analysis
Devise a new severity score based on different patterns of hand movement using sEMG and motion capture analysis | 1 year
  To devise a new severity score based on different patterns of hand movement nursing sEMG and motion capture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ono K, Okada K and Fuji T. Finger escape sign (FES), an objective sign signifying pyramidal tract involvement of the cervical spinal cord. Orthop Trans 1982; 6.2:181.
- [Background] Ono K, Ebara S, Fuji T, Yonenobu K, Fujiwara K, Yamashita K. Myelopathy hand. New clinical signs of cervical cord damage. J Bone Joint Surg Br. 1987 Mar;69(2):215-9. doi: 10.1302/0301-620X.69B2.3818752.
- [Background] Taylor T, Ko S, Mastrangelo C, Bamberg SJ. Forward kinematics using IMU on-body sensor network for mobile analysis of human kinematics. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:1230-3. doi: 10.1109/EMBC.2013.6609729. PMID 24109916